CLINICAL TRIAL: NCT01088932
Title: Phase I, Double-Blind, Placebo-Controlled, Ascending, Multiple-Dose, Safety, Tolerability and Pharmacokinetic Study of SRX246 Capsules in Healthy Adult Volunteers
Brief Title: Multiple Dose Safety Study of SRX246 Capsules in Healthy Volunteers
Acronym: AVN007
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Azevan Pharmaceuticals (Industry)
Responsible Party: Neal G. Simon, PhD, Azevan Pharmaceuticals, Inc.
Allocation: Randomized | Model: Single Group | Masking: Quadruple
Other Study IDs: AVN007
Record Dates: First submitted 2010-03-15; First posted 2010-03-18 (Estimated); Last update posted 2010-07-20 (Estimated); Status verified 2010-07

CONDITIONS: Healthy
Keywords: Safety in Healthy Volunteers
MeSH Terms: interventions — SRX246

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- SRX246 (Experimental): SRX246
  Interventions: Drug: SRX246
- Placebo (Placebo Comparator): placebo
  Interventions: Drug: SRX246

INTERVENTIONS:
Drug: SRX246 — capsules

SUMMARY:
This is a multiple dose clinical study to be conducted with SRX246 capsules to determine the safety, tolerability and pharmacokinetics of the drug over a 14 day dosing period.

DETAILED DESCRIPTION:
This study is intended to evaluate the safety, tolerability and pharmacokinetic profile of multiple oral doses of SRX246 in healthy adult volunteers.

ELIGIBILITY:
Inclusion Criteria:

1. Males and non-pregnant, non-lactating females of non-childbearing potential. Female patients should be either post-menopausal or surgically sterile.
2. Age ≥18 and ≤55 years.
3. Body mass index (BMI) of 18.5 to 34.0 kg/m2, inclusive, and a total body weight of >50kg (110 pounds).
4. In good health as determined by medical history, a baseline physical examination, vital signs, clinical laboratory tests and electrocardiogram (ECG) measurement.
5. Subject is willing and able to sign written informed consent prior to receipt of any study medication or beginning study procedures.
6. Subject is willing and able to follow instructions, comply with the protocol requirements and make all required study visits.

Exclusion Criteria:

1. Pregnant or lactating females, or females of childbearing potential.
2. Subject is positive for HIV, hepatitis B surface antigen or hepatitis C antibody tests at screening.
3. Subject with a positive urine test for drugs of abuse or alcohol at screening or at admission to the clinic on study Day -1.
4. Evidence of any out-of range laboratory value at screening that has not been reviewed, approved and documented as not clinically significant by the Principal Investigator.
5. Subject who has resting supine blood pressure outside of a systolic blood pressure range of 90-140 mmHg or a diastolic blood pressure outside a range of 50-90 mmHg on two consecutive measurements taken up to 10 minutes apart.
6. Subject who has resting supine pulse rate greater than 100 bpm or less than 50 bpm on two consecutive measurements taken up to 10 minutes apart.
7. Subject has taken any alcohol within 48 hours of ANY study-related activities AND cannot abstain from drinking alcohol during the entire duration of the subject's study participation.
8. Subject has used any tobacco products in the past 12 months.
9. A history of significant drug allergy or systemic allergic disease (e.g., urticaria, atopic dermatitis).
10. A general medical or psychological condition or behavior, including current substance dependence or abuse that, in the opinion of the investigator, might not permit the subject to complete the study or sign the informed consent.
11. Any clinically significant abnormality on screening resting 12-lead ECG (e.g., heart block, conduction disorders, ventricular and/or atrial arrhythmias).
12. Any other condition or clinically significant abnormal findings on the physical examination, medical history, or clinical laboratory results during screening that, in the opinion of the Principal Investigator or the Physician Sub-Investigator, would make the subject unsuitable for the study or put them at additional risk.
13. Routine or PRN consumption of medications or herbal supplements that the subject is unable or unwilling to discontinue during the study.
14. Inability to understand or follow study instructions.
15. Treatment with an investigational drug within 30 days preceding the first dose of study medication.
16. Known allergy or hypersensitivity to the investigational study drug/placebo components.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2010-03; Primary Completion 2010-06 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
Safety will be determined by performing vital sign measurements, ECGs, complete physical examinations, hematology and clinical chemistry tests, and recording of any reported adverse experiences. | 14 days

SECONDARY OUTCOMES:
Pharmacokinetics of SRX246 will be determined by taking periodic blood samples for measurement of SRX246 levels. | 14 days

CONTACTS AND LOCATIONS:
Overall Officials: Stephan A Bart, MD, Principal Investigator — SNBL Clinical Pharmacology Center
Locations (1):
- SNBL Clinical Pharmacology Center, Baltimore, Maryland, United States